CLINICAL TRIAL: NCT02852681
Title: A Study to Characterize the Effect of Food on the Bioavailability of 15 mg Estetrol (E4)/3 mg Drospirenone (DRSP) Tablets in Healthy Female Volunteers
Brief Title: Effect of Food on the Bioavailability of 15 mg Estetrol/3 mg Drospirenone Tablets in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Es0001-C101; 2015-001764-19 (EudraCT Number)
Record Dates: First submitted 2016-04-15; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-06

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15 mg E4/3 mg DRSP without food (Other): Treatment A (Reference): a single 15 mg E4/3 mg DRSP tablet without food (fasted).
  Interventions: Drug: 15 mg E4/3 mg DRSP
- 15 mg E4l/3 mg DRSP with food (Other): Treatment B (Test): a single 15 mg E4/3 mg DRSP tablet with food (fed)
  Interventions: Drug: 15 mg E4/3 mg DRSP

INTERVENTIONS:
Drug: 15 mg E4/3 mg DRSP — All subjects received both Treatment A and Treatment B either at the first treatment period (Period 1) or the second treatment period (Period 2). Approximately half of the subjects was randomized to receive either Treatment A followed by Treatment B (Sequence AB), or Treatment B followed by Treatment A (Sequence BA)
  Other Names: 15 mg Estetrol/3 mg Drospirenone

SUMMARY:
This single-center, open-label, randomized, balanced, single-dose, two-treatment, two-period, two-sequence crossover study was conducted under medical supervision in 28 healthy female volunteers.

DETAILED DESCRIPTION:
Food effect bioavailability studies are usually conducted for new drugs and drug products to assess the effect of food on the rate and extent of absorption of a drug when the drug product is administered shortly after a meal (fed conditions), as compared to administration under fasting conditions. Therefore, this study was designed to characterize the effect of a high fat meal on the bioavailability of E4 and DRSP after administration of a single tablet containing 15 mg E4 and 3 mg DRSP.

All subjects entered the study site at least 12 hours before each dosing and fasted for at least 10 hours prior to each dose.

All subjects were to receive both Treatment A (Reference; a single 15 mg E4/3 mg DRSP tablet without food (fasted)) and Treatment B (Test; a single 15 mg E4/3 mg DRSP tablet with food (fed)) either at the first treatment period (Period 1) or the second treatment period (Period 2). Approximately half of the subjects were randomized to receive either Treatment A followed by Treatment B (Sequence AB), or Treatment B followed by Treatment A (Sequence BA).

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy females.
* Between the ages of 18 and 45 years, inclusive.
* Non-smokers who have not used tobacco or nicotine in any form during the 3 months prior to the screening visit.
* Between the body mass index (BMI) of 18 and 30 kg/m2, inclusive, and body weight 45kg.
* Negative serum pregnancy test results at screening and negative urine pregnancy test results before dosing.
* Willing to use double-barrier methods of non-hormonal contraception during the entire study period.

Exclusion Criteria:

Potential study subjects were not entered into and/or may have been discontinued from the study if any of the following applied:

* Use of

  * progestogen-only contraceptive methods [e.g., minipill, implant or, intrauterine system (IUS)] during the last 3 months prior to the first dose or,
  * depot progestogen preparations or an injectable hormonal method of contraception (e.g., Depo-Provera) during the last 6 months prior to the first dose.
* Use (within 28 days prior to first dose) of other hormonal contraceptive method.
* Use of

  * any prescription drugs (except thyroid hormone supplements) or herbal supplements acting on CYP3A4 functions (e.g., St. John's Wort), within 28 days prior to the first dose until study completion,
  * any over-the-counter (OTC) medication (including paracetamol) or dietary supplements (vitamins included) within 14 days prior to the first study dose until study completion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of estetrol in plasma | From day 1 to 4 during both period 1 and period 2
  PK sampling
Cmax of drospirenone in plasma | From day 1 to 4 during both period 1 and period 2
  PK sampling
Area under the plasma concentration versus time curve from time 0 to the last determined concentration (AUC0-tdlc) of estetrol | From day 1 to 4 during both period 1 and period 2
AUC0-tdlc of drospirenone | From day 1 to 4 during both period 1 and period 2
AUC0-inf of estetrol | Day 1 to 4 during both period 1 and period 2
  PK sampling
AUC0-inf of drospirenone | Day 1 to 4 during both period 1 and period 2
  PK sampling

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | From up to day 28 before randomization (28 day screening/run-in period) to day 4 of the Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Dobrin Sviranov, MD, Principal Investigator — Comac Medical

IPD SHARING:
Plan to Share IPD: No